CLINICAL TRIAL: NCT03186690
Title: 154/2013 Grant for Mineral Trioxide Aggregate and Biodentine for Vital Pulp Therapy
Brief Title: Similar Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 154/2013
Record Dates: First submitted 2017-05-27; First posted 2017-06-14 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Deep Caries; Reversible Pulpitis; Irreversible Pulpitis
Keywords: vital pulp therapy; Biodentine; Mineral Trioxide Aggregate
MeSH Terms: interventions — tricalcium silicate; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Intervention Model Description: This prospective longitudinal, parallel-design, randomized clinical trial was set up and is reported according to CONSORT statement
Who Masked: Participant
Masking Description: Participants were not aware of type of capping material used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Experimental): This includes teeth that were treated with Biodntine cement
  Interventions: Other: Biodentine
- Mineral Trioxide Aggregate (Experimental): This includes teeth that were treated with Mineral Trioxide Aggregate (MTA) cement
  Interventions: Other: Mineral Trioxide Aggregate

INTERVENTIONS:
Other: Biodentine
  Arms: Biodentine
Other: Mineral Trioxide Aggregate
  Other Names: MTA
  Arms: Mineral Trioxide Aggregate

SUMMARY:
This study aimed to evaluate the clinical performance of White MTA (MTA, Angelus, Londrina, Brazil) and Biodentine™ in pulp capping of cariously exposed mature permanent teeth.

The investigator performed a prospective longitudinal randomized controlled study utilizing vital permanent mature teeth with deep caries. Patients will be divided randomly into Biodentine™ and MTA groups; Teeth will be assessed clinically and radiographically prior to the procedure. Caries will be excavated under local anesthesia, hemostasis is achieved after pulp exposure using NaOCl and will be capped with Biodentine™ or MTA. Clinical and radiographical follow-up will be performed by a blinded calibrated evaluator after six months and one year, and yearly after.

DETAILED DESCRIPTION:
Study design and ethical approval This prospective longitudinal, parallel-design, randomized clinical trial was set up and is reported according to CONSORT statement. It assessed the outcome of using Biodentine or MTA as a capping material in human mature permanent teeth. Ethical approval for this study was obtained from the Institution Review Board (IRB number (154/13). All participants provided written informed consent after the purpose and methodology were explained in full.

Patient recruitment All patients visiting the Initial Treatment Unit and Post Graduate Dental Clinics were screened for inclusion . Dental examinations were performed to determine whether the patients fulfilled the needed criteria

Approximately 50 subjects will be needed for the study in order to elicit any significant findings as demonstrated by a power analysis from a similar study. The patients will be divided into two groups based on the capping material used. Biodentine™ (Septodont, St. Maur-des-Fossés, France) group, and MTA reparative cement (Angelus, Londrina, Brazil) group. Teeth will be randomly assigned to either group with a coin toss. This included patients with a single offending tooth; the following patient will be then assigned to the other group to keep sample sizes equal in both groups. Patients with more than one offending tooth will have one tooth treated with Biodentine and the other with MTA using again coin toss to randomly distribute capping material among offending teeth.

Clinical examination Pre-operative clinical examinations included a visual inspection of the extent of caries, gingival health, and adjacent soft tissue. A percussion test will be performed, and the periodontal status will be assessed. Pulpal sensibility will also be assessed by cold test with Endo Ice F (Colten-Whaledent, Germany). Patients reporting sharp pain to cold test that did not linger were diagnosed with reversible pulpitis. Patients reporting severe lingering or spontaneous pain were diagnosed with irreversible pulpitis.

Periapical and bitewing radiographs will be obtained for each offending tooth to assess the extent and location of caries, proximity of caries to the pulp, restorability of each tooth, periapical status, and presence of intra-radicular pathosis. Radiographs will be taken using a parallel technique and will be viewed by the naked eye using a viewing box with uniform bright light in a darkened room. All data will be collected by one examiner to ensure reliability.

Clinical protocol Profound local anesthesia of each tooth will achieved by standard infiltration or inferior dental block injection with lidocaine and epinephrine (1:100000) (Xylestesin-A 3M ESPE, Seefeld, Germany). Then, the tooth will be isolated with a rubber dam. The clinical crown disinfected with a cotton pellet soaked in chlorhexidine. Caries will be excavated using a round, high-speed diamond bur with adequate water cooling followed by a round carbide bur. Every attempt will be carried to remove all carious tissue before exposing the pulp. A cotton pellet moistened with 5% NaOCl to be placed into the cavity before pulpal exposure. The size of the pellet varied according to the size of remaining caries; The moistened cotton pellet was left in place for 1-5 minutes to achieve hemostasis. Sodium hypochlorite-soaked cotton will be used to control bleeding in this study.

Once bleeding stopped, capping material will be placed over the exposed pulp. Failure to stop bleeding within additional 3 minutes indicated incomplete removal of the inflamed pulp. In these cases, partial or complete pulpotomy will be performed before capping. Failure to control bleeding after a full pulpotomy indicated propagation of the inflammation to the radicular pulp.

Biodentine™ will be prepared according to the manufacturer's instructions and used to fill half the cavity. Biodentine™ should set within 12 minutes according to the manufacturer. MTA reparative cement will be prepared at a powder:liquid ratio of 3:1 using distilled water according to manufacturer's instructions . MTA to be applied to exposed pulp tissue and adjacent dentine at a thickness of 1.5 to 3 mm. The final restoration will be a resin composite (Z250, 3M, ESPE, USA). Patients are asked to contact the operator if they experience any pain. The first review appointment to be scheduled a week after capping procedure. The patient will be questioned about sensitivity, mastication discomfort, and sensations of pain.

Recall protocol Six-month and yearly after follow-up appointments will be scheduled. Patients, who are not aware of the type of capping material received, will be questioned about pain, sensitivity, and mastication discomfort. Clinical examinations to be performed to detect soft tissue swelling, sinus tract, the integrity of the coronal restoration, and tooth mobility. The review visits to be performed blindly by another operator. Radiographical examinations will also be performed to evaluate the periapical status, the formation of the dentine bridge, pulpal calcifications, or canal obliteration and evidence of tooth discoloration. Tooth vitality will be monitored by cold tests. Treatment was considered successful based on the following features: absence of severe spontaneous pain, no discomfort while eating, no soft tissue swelling, mobility that is no greater than grade I, the absence of periapical rarefaction, internal or external resorption, root canal obliteration, and normal viability following pulpotomy.

Statistical analysis The data will be processed using the JMP software (SAS Institute Inc., North Carolina, United States) with alpha=0.05. The chi-square test (significance level of < 0.05) will be used to determine differences between the success rates of Biodentine and MTA. The survival probabilities will be compared using The Wilcoxon and the log-rank tests.

ELIGIBILITY:
Inclusion Criteria:

* Teeth that Fulfilled All the Following Criteria Were Selected
* Vital teeth responding positively to cold test.
* Reversible or irreversible pulpitis with or without periapical lesion.
* Deep caries that if removed exposure of the pulp is most likely to occur.
* Permanent mature molar, premolar or anterior tooth
* The tooth should be restorable.
* No serious medical problem that could prevent the patient from receiving the treatment or attending later the follow up visits.

Exclusion Criteria:

* Exclusion Criteria
* Immature tooth
* Unrestorable tooth
* Tooth that did not respond to cold test
* Serious medical problem that could prevent the patient from receiving the treatment or attending later the follow up visits.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2023-10-04 (Estimated)

PRIMARY OUTCOMES:
clinical vital pulp therapy success | from date of randomization until failure reported for up to 100 months
  Treatment was considered successful based on absence of symptoms and signs

SECONDARY OUTCOMES:
Radiographic success | from date of randomization until failure reported for up to 100 months
  treatment could be further evaluated based on absence of canal oblitration

CONTACTS AND LOCATIONS:
Overall Officials: Lama Awawdeh, PhD, Study Chair — Jordan University of Science and Technology
Locations (1):
- Dr Lama Awawdeh, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No